CLINICAL TRIAL: NCT02747290
Title: Safety and Diagnostic Performance of 68Gallium-labeled NOTA-BBN-RGD PET/CT in Prostate Cancer Patients
Brief Title: 68Ga-NOTA-BBN-RGD PET/CT in Prostate Cancer Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCHNM011; ZIAEB000073 (NIH)
Record Dates: First submitted 2016-04-19; First posted 2016-04-21 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-03

CONDITIONS: Prostate Cancer
Keywords: BBN-RGD; PET; integrin αvβ3; GRPR
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 68Ga-NOTA-BBN-RGD PET/CT (Experimental): The patients were injected with 111-148 MBq of 68Ga-NOTA-BBN-RGD in one dose intravenously and underwent PET/CT scan 15-30 min later.
  Interventions: Drug: 68Ga-NOTA-BBN-RGD

INTERVENTIONS:
Drug: 68Ga-NOTA-BBN-RGD — 68Ga-NOTA-BBN-RGD were injected into the patients before the PET/CT scans

SUMMARY:
This is an open-label positron emission tomography/computed tomography (PET/CT) study to investigate the diagnostic performance and evaluation efficacy of 68Ga-NOTA-BBN-RGD in prostate cancer patients. A single dose of 111-148 Mega-Becquerel (MBq) 68Ga-NOTA-BBN-RGD will be injected intravenously. Visual and semiquantitative method will be used to assess the PET/CT images.

DETAILED DESCRIPTION:
Both GRPR and integrin αvβ3 are overexpressed in neoplastic cells of human prostate cancer. To target both receptors, a heterodimeric peptide BBN-RGD was synthesized from bombesin(7-14) and c(RGDyK) through a glutamate linker and then labeled with 68Ga. An open-label whole-body PET/ CT study was designed to investigate the safety and dosimetry of 68Ga-NOTA-BBN-RGD and diagnostic performance of 68Ga-NOTA-BBN-RGD PET/CT in patients with primary and/or metastasis prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to provide a written informed consent, needle biopsy diagnosed as prostate cancer, have undergone whole body bone scan, able to provide basic information and sign the written informed consent.

Exclusion Criteria:

* The exclusion criteria included claustrophobia, kidney or liver failure, and inability to fulfill the study.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value of 68Ga-NOTA-BBN-RGD in prostate cancer | 1 year
  The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake value (SUV) of the tracer in prostate cancer will be measured.

SECONDARY OUTCOMES:
Adverse events collection | 1 week
  Adverse events within 1 week after the injection and scanning of patients and patients will be followed and assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Li, MD., Study Chair — Peking Union Medical College Hospital, Chinese Academy of Medical Science and Peking Union Medical College
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China